CLINICAL TRIAL: NCT02573896
Title: A Phase I Dose Escalation Study of Autologous Expanded Natural Killer (NK) Cells for Immunotherapy of Relapsed Refractory Neuroblastoma With Dinutuximab +/- Lenalidomide
Brief Title: Immunotherapy of Relapsed Refractory Neuroblastoma With Expanded NK Cells
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: New Approaches to Neuroblastoma Therapy Consortium (Other)
Collaborators: Nationwide Children's Hospital (Other); United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NANT 2013-01
Record Dates: First submitted 2015-09-16; First posted 2015-10-12 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Neuroblastoma
Keywords: relapsed refractory neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — dinutuximab; IL32 protein, human; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NK cells with Dinutuximab & Lenalidomide (Experimental): Patients in this arm will receive a designated dose of NK cells on Day 5 and 17.5 mg/m2/dose of dinutuximab on Day 1-4. Patients on Dose Level 4 will also receive 25mg/m2/dose of Lenalidomide during Day -6 through 14 of treatment.
  Interventions: Drug: Dinutuximab; Biological: NK Cells; Drug: Lenalidomide

INTERVENTIONS:
Drug: Dinutuximab — 17.5 mg/m2/day of dinutuximab will be given for 4 consecutive days (days 1-4 of each course) via intravenous infusion over ten hours.
  Other Names: Chimeric Monoclonal Antibody 14.18; MAB Ch 14.18; Unituxin
Biological: NK Cells — The designated dose of NK Cells will be infused on Day 5 by IV drip using a Y infusion set with a filter-less chamber. Cells should not be delivered at a rate faster than 10 ml/kg/hr (as determined by drip rate or syringe push rate), and should not take longer than one hour for total infusion time if possible.
  Other Names: Natural Killer Cells
Drug: Lenalidomide — 25 mg/m2/day of Lenalidomide will be given at Dose Level 4, once daily with or without food by mouth on days -6 through +14.

SUMMARY:
This NANT trial will determine the maximum tolerated dose (MTD) of autologous expanded natural killer (NK) cells when combined with standard dosing of dinutuximab and will assess the feasibility of adding lenalidomide at the recommended Phase II dose of the expanded NK cells with dinutuximab, for treatment of children with refractory or recurrent neuroblastoma.

DETAILED DESCRIPTION:
This NANT trial will determine the maximum tolerated dose (MTD) of autologous expanded natural killer (NK) cells when combined with standard dosing of dinutuximab and will assess the feasibility of adding lenalidomide at the recommended Phase II dose of the expanded NK cells with dinutuximab, for treatment of children with refractory or recurrent neuroblastoma.

Dinutuximab is a chimeric antibody against GD2, which is expressed on a majority of neuroblastoma cells. It has been shown to increase EFS and OS in patients with high-risk neuroblastoma when given after autologous stem cell transplant in combination with subcutaneous GM-CSF and intravenous IL-2, followed by isotretinoin. Lenalidomide has been studied in children with solid tumors and can safely be given to patients based on 2 prior trials in children. It was also shown to have immunomodulatory effects and is synergistic with dinutuximab. Lenalidomide is also an oral agent that can be given in the outpatient setting. Natural killer cells are lymphocytes of the innate immune system that have the ability to recognize and kill malignant cells, including neuroblastoma. Dinutuximab and lenalidomide both exert part of their anti-cancer effect through the activation of natural killer cells. Patients were given these in combination in the NANT 2011-04 study where the safety and immunomodulatory effect were established. The dose level proposed in this study is based off of these data. Natural killer cells are dysfunctional and low in number in many cancer patients, and number and function are further suppressed by chemotherapy and radiation. Investigators hypothesize that autologous NK cells can be expanded and activated ex vivo and readministered to restore number and function, and in combination with lenalidomide and dinutuximab will provide an anti-tumor effect in patients with relapsed or refractory neuroblastoma.

Investigators will determine the feasibility of centralized expansion, cryopreservation, and distribution of autologous NK cells. Investigators will then determine the maximum tolerated dose by assessing the toxicities of autologous expanded NK cells given with dinutuximab; by assessing the toxicities, cytokinetics and immunomodulatory effects, Investigators will select the recommended Phase II dose of the two-agent combination after dose escalation of the NK cells and then adding lenalidomide to the combination to establish the three-agent combination.

Cytokinetics (persistence of infused NK cells) and immune function studies will be required for all patients entered on this study. In addition to routine assessment of response, quantification of rare tumor cell detection in blood and bone marrow using TLDA will also provide another measure of possible anti-tumor efficacy to support the rationale for the final schedule chosen.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be less than or equal to 30 years of age when registered on study
2. Patients must have a diagnosis of neuroblastoma either by histologic verification of neuroblastoma and/or demonstration of tumor cells in the bone marrow with increased urinary catecholamines.
3. Patients must have a history of high-risk neuroblastoma according to COG risk classification at the time of study registration. Patients who were initially considered low or intermediate-risk, but then reclassified as high-risk are also eligible.
4. All patients must have at least one of the following

   a) Recurrent/progressive disease: after the diagnosis of high risk neuroblastoma at any time prior to enrollment regardless of response to frontline therapy b) No prior history of recurrent/progressive disease since the diagnosis of high risk neuroblastoma b1) Refractory disease- a best overall response of no response/stable disease since diagnosis of high risk neuroblastoma and at least 4 cycles of induction therapy. No prior history of recurrent/progressive disease since the diagnosis of high risk neuroblastoma.

   b2) Persistent disease- a best overall response of no partial response since diagnosis of high risk neuroblastoma and at least 4 cycles of induction therapy. No prior history of recurrent/progressive disease since the diagnosis of high risk neuroblastoma.
5. Patients must have at least ONE of the following (lesions may have received prior radiation therapy as long as they meet the other criteria listed below):

   1. For recurrent/progressive or refractory disease, at least one MIBG avid bone site.
   2. For persistent disease, if a patient has 3 or more MIBG avid lesions, then no biopsy is required. If a patients has only 1 or 2 MIBG avid bone lesion sites then biopsy confirmation of neuroblastoma or ganglioneuroblastoma in at least one MIBG avid site present at the time of enrollment is required to be obtained at any time point prior to enrollment.
   3. For MIBG non-avid tumors, patients must have at least one FDG avid site and a biopsy confirmation of neuroblastoma and/or ganglioneuroblastoma at any time prior to enrollment from at least one FDG-avid site.
6. Any amount of neuroblastoma tumor cells in the bone marrow done at the time of study enrollment based on routine morphology with or without immunocytochemistry in at least one sample from bilateral aspirates and biopsies.
7. At least one soft tissue lesion that meets criteria for a TARGET lesion as defined by:

   1. SIZE: Lesion can be accurately measured in at least one dimension with a longest diameter ≥ 10 mm, or for lymph nodes ≥ 15 mm on short axis. Lesions meeting size criteria will be considered measurable.
   2. In addition to size, a lesion needs to meet one of the following criteria except for patients with parenchymal CNS lesions which only need to meet size criteria:

   b1) MIBG avid. For patients with recurrent/progressive or refractory disease, no biopsy is required. For patients with persistent disease only: If a patient has only 1 or 2 MIBG avid lesions sites, then biopsy confirmation of neuroblastoma and/or ganglioneuroblastoma in at least one MIBG avid site present at time of enrollment is required to be obtained. If a patient has 3 or more MIBG avid lesions, then no biopsy is required.

   b2) MIBG non avid tumors: Patients must have at least one FDG avid site and biopsy confirmation of neuroblastoma and/or ganglioneuroblastoma in at least one FDG-PET avid site present at the time of enrollment.
8. At least one non-target soft tissue lesion that is not measurable, but had a biopsy positive for neuroblastoma and/or ganglioneuroblastoma or is MIBG avid at any time prior to enrollment.
9. Patients must have a life expectancy of at least 12 weeks and a Lansky (≤16 years) or Karnofsky (>16 years) score of at least 50.
10. Prior Therapy 1. Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to study registration.

2. Patients must not have received the therapies indicated below after disease evaluation or within the specified time period prior to registration on this study as follows:

1. Myelosuppressive chemotherapy: must not have received within 2 weeks prior to registration.
2. Biologic anti-neoplastics- agents not known to be associated with reduced platelet or ANC counts (including retinoids): must not have received within 7 days prior to registration.
3. Monoclonal antibodies: must have received last dose at least 7 days or 3 half-lives whichever is longer, but no longer than 30 days (with recovery of any associated toxicities), prior to protocol therapy.
4. Cellular Therapy (e.g. modified T cells, NK cells, dentritic cells etc.):

   must not have received within 3 weeks and resolution of all toxicities.
5. Radiation: must not have received small port radiation within 7 days prior to registration.
6. Hematopoietic Stem Cell Transplant:
7. IVIG

11) All patients must have adequate organ function defined as:

- Hematological Function:

1. Absolute Phagocyte count (APC= neutrophils and monocytes): ≥ 1000/µL
2. Absolute Neutrophil count: ≥750/µL
3. Absolute Lymphocyte count ≥ 500/µL
4. Platelet count: ≥ 50,000/µL, transfusion independent (no platelet transfusions within 1 week)
5. Hemoglobin ≥ 10 g/dL (may transfuse)
6. Patients with known bone marrow metastatic disease will be eligible for study as long as they meet hematologic function criteria above.

   * Renal Function: Age-adjusted serum creatinine ≤ to 1.5 x normal for age/gender OR creatinine clearance or GFR greater than or equal to 60 cc/min/1.73m2
   * Liver Function: Total bilirubin ≤ 1.5 x normal for age, AND SGPT (ALT) 135 and SGOT (AST) ≤ 3 x upper limit of normal. Sinusoidal obstruction syndrome (SOS) if present, must be stable or improving clinically
   * Cardiac Function: Normal ejection fraction documented by either echocardiogram or radionuclide MUGA evaluation OR Normal fractional shortening documented by echocardiogram
   * Pulmonary Function: No dyspnea at rest, no oxygen requirement.

     12) Reproductive Status: All post-menarchal females must have a negative beta-HCG. Males and females of reproductive age and childbearing potential must use effective contraception for the duration of their participation.

     13) Patients with other ongoing serious medical issues must be approved by the study chairprior to registration.

     14) Patients may not receive any other anti-cancer agents or radiotherapy while on protocol therapy.

     15) Ability to Swallow Pills

Exclusion Criteria:

1. Pregnancy: Quantitative Serum B-HCG must be negative in girls who are post-menarchal.
2. Breast feeding women are not eligible.
3. Active or uncontrolled infection
4. CNS metastasis.
5. Hypersensitivity to thalidomide, including history of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs (dose level 4 only).
6. Patient declines participation in NANT 2004-05; unless the institution has been granted special exemption from mandatory registration on NANT 2004-05 by the NANT Operations Center.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
NK cell production feasibility (lowest dose level) | After cell expansion, day 4 of protocol therapy
  Proportion of patients whose NK cell product is at least 80% of 10^7 NK cells per kg (sufficient cells to give at least 1 dose at the lowest dose level).
NK cell production feasibility | After cell expansion, day 4 of protocol therapy
  Proportion of patients whose NK cell product is at least 80% of the planned dose for one dose
MTD/RP2D determination | all toxicities from enrollment through 30 days following end of protocol therapy
  Proportion of patients with any Grade 3 or greater non-hematological toxicities on any course

SECONDARY OUTCOMES:
Describe Non-Hematological Toxicities | all toxicities from enrollment through 30 days following end of protocol therapy
  Proportion of patients with any Grade 3 or greater non-hematological toxicities on any course
Describe Hematological Toxicities | all toxicities from enrollment through 30 days following end of protocol therapy
  Proportion of patients with any Grade 3 or greater hematological toxicities on any course
Overall Response | From Day 1 of protocol therapy through 30 days following end of protocol therapy
  Proportion of patients evaluable for response with a best overall response of CR/CR-MD/PR

CONTACTS AND LOCATIONS:
Overall Officials: Araz Marachelian, MD, MS, Study Chair — Children's Hospital Los Angeles
Locations (11):
- United States (11):
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - University of Chicago Comer Children's Hospital, Chicago, Illinois
  - Childrens Hospital Boston, Dana-Farber Cancer Institute., Boston, Massachusetts
  - C.S Mott Children's Hospital, Ann Arbor, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cook Children's Healthcare System, Fort Worth, Texas
  - Seattle Children's Hospital, Seattle, Washington